CLINICAL TRIAL: NCT05277571
Title: A Phase 1/2A, Randomized, Placebo-Controlled, Single-Ascending Dose (Part A, Participant- and Investigator-Blind) and Repeat-Dose (Part B, Participant-, Investigator-, and Sponsor-Blind) Study to Investigate the Safety, Pharmacokinetics, and Efficacy (Part B Only) of UCB1381 in Healthy Study Participants (Part A) and in Study Participants With Moderate to Severe Atopic Dermatitis (Part B)
Brief Title: A Single-ascending Dose (Part A) and Repeat-dose (Part B) Study to Investigate the Safety, Pharmacokinetics and Efficacy (Part B Only) of UCB1381 in Healthy Study Participants (Part A) and in Study Participants With Moderate to Severe Atopic Dermatitis (Part B)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0110
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Phase 1/2A; Healthy study participants; Patients; UCB1381
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- UCB1381 dosing regime 1 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 intravenously (iv).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 2 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 intravenously (iv).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 3 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 intravenously (iv).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 4 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 intravenously (iv).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 5 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 subcutaneously (sc).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 6 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 subcutaneously (sc).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 7 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 intravenously (iv).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 8 in Part A (Experimental): Participants will be randomized to receive a single dose UCB1381 intravenously (iv).
  Interventions: Biological: UCB1381
- UCB1381 dosing regime 9 in Part B (Experimental): Participants will be randomized to receive repeated doses UCB1381 intravenously (iv).
  Interventions: Biological: UCB1381
- Placebo iv Arm Part A (Placebo Comparator): Participants will be randomized to receive a single dose of placebo iv to maintain the blinding.
  Interventions: Drug: Placebo
- Placebo sc Arm Part A (Placebo Comparator): Participants will be randomized to receive a single dose of placebo sc to maintain the blinding.
  Interventions: Drug: Placebo
- Placebo iv Arm Part B (Placebo Comparator): Participants will be randomized to receive repeated doses of placebo iv to maintain the blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: UCB1381 — UCB1381 will be administered intravenously (iv) or subcutaneously (sc) in different dosages in Part A and iv in Part B
  Arms: UCB1381 dosing regime 1 in Part A; UCB1381 dosing regime 2 in Part A; UCB1381 dosing regime 3 in Part A; UCB1381 dosing regime 4 in Part A; UCB1381 dosing regime 5 in Part A; UCB1381 dosing regime 6 in Part A; UCB1381 dosing regime 7 in Part A; UCB1381 dosing regime 8 in Part A; UCB1381 dosing regime 9 in Part B
Drug: Placebo — Placebo will be administered iv or sc in Part A and iv in Part B to maintain the blinding.
  Arms: Placebo iv Arm Part A; Placebo iv Arm Part B; Placebo sc Arm Part A

SUMMARY:
The purpose of the study is to investigate the safety and tolerability of single-ascending doses of UCB1381 (intravenous and subcutaneous) in healthy study participants and after repeat intravenous dosing in study participants with atopic dermatitis. Efficacy will be assessed following repeat intravenous dosing versus placebo in study participants with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

Part A Healthy study participants

* Participant must be 18 to 55 years of age inclusive at the time of signing the informed consent form (ICF)
* Participant must be overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participant has a body mass index (BMI) within the range 18 to 30 kg/m2 (inclusive)
* Participant can be male or female and must agree to use contraception

Part B Participants with moderate to severe Atopic dermatitis (AtD)

* Participant must be 18 to 65 years of age inclusive at the time of signing the ICF
* Participant has moderate or severe AtD that has been present for at least 12 months prior to initiating the study (signing of the ICF) and with:
* A validated Investigator Global Assessment (vIGA) score ≥3 at Screening and Baseline
* An Eczema Area and Severity Index (EASI) score of ≥14 at Screening and ≥16 at Baseline
* Pruritis Numerical Rating Scale (NRS) ≥3 at Screening and Baseline
* ≥10 % body surface area (BSA) of AtD involvement at Screening and Baseline
* Either documented recent history (within 6 months before the Screening Visit) of inadequate response to treatment with topical medications (regular use of topical corticosteroids [TCS] or topical calcineurin inhibitors [TCIs]) or when topical treatments are confirmed to be otherwise medically inadvisable (eg, because of important side effects or safety risks)
* Participant has a BMI within the range 18 to 35 kg/m2 (inclusive)

Exclusion Criteria:

Part A Healthy study participants

* Participant has a history or presence of any medical or psychiatric condition, physical examination finding, laboratory test result, electrocardiogram (ECG), or vital sign that, in the opinion of the investigator, could significantly alter the absorption, metabolism, or elimination of drugs; constitute a risk when taking the study intervention; or interfere with the interpretation of data
* Participant has a known hypersensitivity to any components of the investigational medicinal product (IMP) or other biologic drugs (including humanized monoclonal antibodies (mAbs)), clinically significant drug allergies, or history of severe adverse reactions after drug administration
* Participant has a past history of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis)
* Participant has previously been randomized in this study
* Participant has participated in another study of an IMP or has received any biologic agent (such as mAbs, including marketed drugs and including biologic agents that target interleukin (IL)-13 or IL-22) within the 30 days prior to Screening or 5 half-lives (whichever is longer), if this information can be validated by the investigator

Part B Participants with moderate to severe AtD

* Participant has a history or presence of any medical or psychiatric condition, physical examination finding, laboratory test result, electrocardiogram (ECG), or vital sign that, in the opinion of the investigator, could significantly alter the absorption, metabolism, or elimination of drugs; constitute a risk when taking the study intervention; or interfere with the interpretation of data
* Participant has a known hypersensitivity to any components of the IMP or other biologic drugs (including humanized mAbs), clinically significant drug allergies, or history of severe adverse reactions after drug administration
* Participant has a past history of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis)
* Participant has had pharmaceutically active topical therapies for AtD (including mild topical corticosteroids (TCS)) within 2 weeks of the Baseline Visit (corticosteroids, cyclosporin or other calcineurin inhibitors [eg, tacrolimus, pimecrolimus])
* Participant has received phototherapy or systemic non-biologic therapies for AtD within 4 weeks of the Baseline Visit (including moderate/strong corticosteroids, cyclosporine A or other calcineurin inhibitors, mycophenolate mofetil, azathioprine, methotrexate, or any alternative medicine for AtD, eg, traditional Chinese medicine)
* Participant has previously used a biologic that affects IL-13 or IL-22 pathways, or any JAK inhibitor (including marketed and/or experimental treatments), within 30 days or 5 half-lives (whichever is longer) of the Baseline Visit. Previous use of biologics affecting IL-13 or IL-22 pathways is only accepted if treatment was stopped due to reasons other than inadequate efficacy and safety (eg, administrative reasons, poor convenience, poor access to drug)
* Participant has received any prescription or nonprescription medicines, including over the counter remedies and herbal and dietary supplements (other than vitamins within recommended daily dose limits) within 14 days (or 5 half-lives of the respective drug, whichever is longer) prior to the Baseline Visit, other than contraceptives (oral, implant, or intrauterine devices) or occasional use of analgesics such as paracetamol (acetaminophen, with or without caffeine, with a maximal dose of 4g/day and 10g/14 days) or intranasal corticosteroids for seasonal rhinitis or inhaled bronchodilators and low dose inhaled corticosteroids for mild asthma. In case of uncertainty, the UCB Development Physician should be consulted
* Participant has previously been randomized in this study
* Participant has participated in previous studies with a biologic that affects IL-13 or IL-22 pathways, or any JAK inhibitor (including marketed and/or experimental treatments), within 30 days or 5 half-lives (whichever is longer) of the Baseline Visit. Previous use of biologics affecting IL-13 or IL-22 pathways is only accepted if treatment was stopped due to reasons other than inadequate efficacy and safety (eg, administrative reasons, poor convenience, poor access to drug)
* Participant has participated in another study of an IMP within 30 days or 5 half-lives (whichever is longer) of the Baseline Visit or is currently participating in another study of an IMP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Incidents of treatment-emergent adverse events (TEAEs) from Baseline through the End of Study (EOS) Visit (Week 12) in Part A | From Baseline up to Week 12 in Part A
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study medication.
Incidents of treatment-emergent serious adverse events (TESAEs) from Baseline through the EOS Visit (Week 12) in Part A | From Baseline up to Week 12 in Part A
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Incidents of TEAEs from Baseline through the EOS Visit (Week 22) in Part B | From Baseline up to Week 22 in Part B
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study medication.
Incidents of TESAEs from Baseline through the EOS Visit (Week 22) in Part B | From Baseline up to Week 22 in Part B
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
≥75% improvement vs Baseline (Yes/No) in Eczema Area and Severity Index score (EASI75) at Week 12 in Part B | From Baseline up to Week 12 in Part B
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema. A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.

SECONDARY OUTCOMES:
UCB1381 Cmax from Baseline through the EOS Visit (Week 12) in Part A | From Baseline up to Week 12 in Part A
  Cmax: Maximum observed concentration
UCB1381 Tmax from Baseline through the EOS Visit (Week 12) in Part A | From Baseline up to Week 12 in Part A
  Tmax: Time of observed Cmax
UCB1381 AUC(0-t) from Baseline through the EOS Visit (Week 12) in Part A | From Baseline up to Week 12 in Part A
  AUC(0-t): Area under the concentration-time curve from time zero to the time of last detectable concentration.
UCB1381 AUC from Baseline through the EOS Visit (Week 12) in Part A | From Baseline up to Week 12 in Part A
  AUC: Area under the concentration-time curve from time zero to infinity.
UCB1381 F% from Baseline through the EOS Visit (Week 12) in Part A | From Baseline up to Week 12 in Part A
  F%: Bioavailability of subcutaneous administration
Percent change from Baseline in EASI score at Week 12 in Part B | From Baseline up to Week 12 in Part B
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema. A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.
≥50% improvements vs Baseline (Yes/No) in EASI score (EASI50) at Week 12 in Part B | From Baseline up to Week 12 in Part B
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema. A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.
≥90% improvements vs Baseline (Y/N) in EASI score (EASI90) at Week 12 in Part B | From Baseline up to Week 12 in Part B
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema. A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.
Validated Investigator Global Assessment (vIGA) score of 0 or 1 (Y/N) at Week 12 in Part B | From Baseline up to Week 12 in Part B
  vIGA: Validated Investigator Global Assessment score is using descriptors that best describe the overall appearance of the lesions at a given time point. Assessment: vIGA 0=clear, vIGA 1=almost clear, vIGA 2=mild, vIGA 3=moderate, vIGA 4=severe
UCB1381 Cmax at week 12 after the final dose in Part B | From Baseline up to Week 12 in Part B
  Cmax: Maximum observed concentration
UCB1381 Tmax at week 12 after the final dose in Part B | From Baseline up to Week 12 in Part B
  Tmax: Time of observed Cmax
UCB1381 AUCtau at week 12 after the final dose in Part B | From Baseline up to Week 12 in Part B
  AUCtau: Area under the curve for the dosing interval after the final dose.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (16):
- United States (16):
  - Up0110 125, Beverly Hills, California
  - Up0110 101, Glendale, California
  - Up0110 116, Los Angeles, California
  - Up0110 121, Northridge, California
  - Up0110 126, Tustin, California
  - Up0110 127, Valencia, California
  - Up0110 108, Clearwater, Florida
  - Up0110 109, Miami Lakes, Florida
  - Up0110 106, Ocala, Florida
  - Up0110 102, St. Petersburg, Florida
  - Up0110 111, College Park, Georgia
  - Up0110 114, Minneapolis, Minnesota
  - Up0110 107, New York, New York
  - Up0110 124, Winston-Salem, North Carolina
  - Up0110 104, Oklahoma City, Oklahoma
  - Up0110 119, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of reidentifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org